CLINICAL TRIAL: NCT02724683
Title: Management of Symptomatic Malignant Ascites With an Patient-controlled, Vascular Catheter - a Validation Study.
Brief Title: Symptomatic Ascites Drainage With a Patient-controlled Vascular Catheter.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maciej Stukan, MD, PhD (Other Government)
Responsible Party: Sponsor-Investigator, Maciej Stukan, MD, PhD, Dr, Gdynia Oncology Center
Organization: Gdynia Oncology Center (Other Government)
Other Study IDs: GCO-1
Record Dates: First submitted 2016-03-20; First posted 2016-03-31 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Malignant Ascites
Keywords: ascites; drainage; catheter; symptoms; management; quality of life; malignant; cancer
MeSH Terms: conditions — Ascites; Neoplasms | interventions — Vascular Access Devices; Interviews as Topic; Quality of Life; Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptomatic ascites drainage with CVC.: Patients with malignant, symptomatic, refractory ascites. Ascites drainage with vascular catheter (CVC) inserted into abdominal cavity will be performed. Patients will be asked to complete interview, quality of life questionnaire, nutritional status assessment and quality of procedure survey.
  Interventions: Device: Ascites drainage with vascular catheter.; Behavioral: Interview.; Behavioral: Quality of life.; Device: Quality of procedure.; Other: Nutritional status

INTERVENTIONS:
Device: Ascites drainage with vascular catheter. — In case of symptomatic malignant ascites, the procedure of vascular catheter insertion into abdominal cavity will be performed, followed by slow, systematic drainage, on patient's demand.
Behavioral: Interview. — Interview with patients will be performed according to attached chart. The aim is to collect data concerning patient's symptoms, co-morbidity, and basic clinical data about the primary malignancy and treatment status.
Behavioral: Quality of life. — Quality of life questionnaire (QLQ). Patients will be asked to complete QLQ at two time points: 1. immediately before the procedure, 2. one or two weeks after the procedure.
Device: Quality of procedure. — Patients will be asked to complete quality of procedure questionnaire at one time point: one or two weeks after the procedure.
Other: Nutritional status — Risk of malnutrition and ability to feed normally will be assessed with specific questionnaire at two time points: 1. immediately before the procedure, 2. one or two weeks after the procedure.

SUMMARY:
The purpose of this study is to determine whether drainage with the usage of a fine, patient-controlled vascular catheter inserted into abdominal cavity is a feasible, safe and effective method in the management of symptomatic malignant ascites. Complications' rate of the procedure and patients' quality of life, nutritional status and experience on the treatment are main endpoints.

DETAILED DESCRIPTION:
Patients with symptomatic, refractory malignant ascites (MA) will be eligible for the study. In case a cancer treatment is not effective against ascites, or no target, systemic treatment is possible patients will be eligible for percutaneous placement of a vascular catheter into abdominal cavity followed be drainage performed in a regular basis when required, at home or ambulatory. Adult patients with every malignant disease, female and male, and coexisting symptomatic MA can be recruited.

Clinical, quality of life (QOL) and quality of the procedure data will be collected. The study is planned to be a multiinstitutional. A template is provided to collect essential clinical data concerned with a patient, malignant disease, procedure performance and complications. QOL and patients' experience on the treatment is to be evaluated with formal questionnaires - EORTC C15-PAL and FACIT-TS-G - permission to use granted from EORTC and FACIT respectively. Additionally, a nutrition monitoring will be performed (if possible and feasible) in patients with MA and drainage.

Data will be saved in a computer, secured data base for calculations. A cohort of 150 patients is planned to be collected. Duration of the study will depend on how many institutions will participate, and how fast patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic, refractory malignant ascites,
* supportive care (professional or family members) available at patients' home,
* informed signed consent of the patient.

Exclusion Criteria:

* ascites not of malignant origin,
* asymptomatic ascites,
* suspected or clinically apparent infection especially at the site of planned drainage placement,
* significant coagulopathy,
* very poor performance status (PS4),
* patient not able to read and sign informed consent,
* mucinous ascites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients considered eligible are those with malignant disease of any origin and coexisting symptomatic ascites who require a management anyway.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2016-01; Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events. | 2 weeks
  Early and late adverse events of the catheter placement and later drainage to be recorded.
Change in quality of life. | 2 weeks
  Change in quality of life measured with standard questionnaire EORTC-C15-PAL before the procedure and 1-2 weeks later.

SECONDARY OUTCOMES:
Number of participants with drainage complication during cancer treatment vs observation. | 1 month
  Assessment of possibilities to provide cancer treatment with active ascites drainage via catheter, by reporting number of participants with adverse events during chemotherapy or radiotherapy, whichever applies and comparison to observation (patients with palliative intent only, no active cancer treatment).
Number of participants with successful catheter placement. | 2 weeks
  From all eligible participants a number of participants with successful catheter placement followed by effective drainage will be recorded.
Patient's experience on the treatment. | 2 weeks
  Patient's experience on the treatment measured with standard questionnaire (FACIT-TS-G).
Change in nutrition habits. | 2 weeks
  Changes in ability to feed assessed in a descriptive way with the Subjective Global Assessment (SGA) questionnaire.

OTHER OUTCOMES:
Change in nutrition status among participants with prolonged ascites drainage. | 1 month
  Risk of malnutrition and ability to feed normally to be assessed with Subjective Global Assessment (SGA) questionnaire among participants with prolonged (1-2 months) ascites drainage.
Number of ambulatory visits or hospital admissions. | 1 month
  Number of ambulatory visits or hospital admissions to manage symptoms caused by ascites.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Stukan, MD, Principal Investigator — Gdynia Oncology Center
Locations (2):
- The Central and Eastern European Gynecologic Oncology Group (CEEGOG), Prague, Czechia
- Gdynia Oncology Center, Gdynia, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hui D, Bruera E. Integrating palliative care into the trajectory of cancer care. Nat Rev Clin Oncol. 2016 Mar;13(3):159-71. doi: 10.1038/nrclinonc.2015.201. Epub 2015 Nov 24. PMID 26598947
- [Result] Stephenson J, Gilbert J. The development of clinical guidelines on paracentesis for ascites related to malignancy. Palliat Med. 2002 May;16(3):213-8. doi: 10.1191/0269216302pm509oa. PMID 12046997
- [Result] Becker G, Galandi D, Blum HE. Malignant ascites: systematic review and guideline for treatment. Eur J Cancer. 2006 Mar;42(5):589-97. doi: 10.1016/j.ejca.2005.11.018. Epub 2006 Jan 24. PMID 16434188
- [Result] Stukan M, Lesniewski-Kmak K, Wroblewska M, Dudziak M. Management of symptomatic ascites and post-operative lymphocysts with an easy-to-use, patient-controlled, vascular catheter. Gynecol Oncol. 2015 Mar;136(3):466-71. doi: 10.1016/j.ygyno.2014.11.073. Epub 2014 Nov 28. PMID 25434633
- [Result] da Silva Fink J, Daniel de Mello P, Daniel de Mello E. Subjective global assessment of nutritional status - A systematic review of the literature. Clin Nutr. 2015 Oct;34(5):785-92. doi: 10.1016/j.clnu.2014.12.014. Epub 2014 Dec 26. PMID 25596153
- [Result] Stukan M. Drainage of malignant ascites: patient selection and perspectives. Cancer Manag Res. 2017 Apr 12;9:115-130. doi: 10.2147/CMAR.S100210. eCollection 2017. PMID 28442933